CLINICAL TRIAL: NCT04492813
Title: Comparison of Plasmatic Concentrations of Propofol and Remifentanil During Monitored Anesthesia in Obese and Non Obese Patients.
Brief Title: Plasmatic Concentrations of Propofol and Remifentanil in Obese and Non Obese Patients.
Acronym: COCOPOPONO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: COCOPOPONO
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: General Anesthesia; Obesity
Keywords: General anesthesia; Obesity; Propofol pharmacokinetic; Remifentanyl pharmacokinetic
MeSH Terms: conditions — Obesity | interventions — Remifentanil

STUDY DESIGN:
Intervention Model Description: Each obese patient is matched with a non-obese patient by considering a pairing according to age (more or less 5 years), gender and renal function (more or less 10ml / min / 1.73m² creatinine clearance).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obese patients (Experimental): Severe and morbidly obese patients (35²≤BMI <55)
  Interventions: Drug: Pharmacokinetic of propofol and remifentanil
- Non Obese patients (Active Comparator): Patients with normal weight or slightly overweight (19 <BMI <30).
  Interventions: Drug: Pharmacokinetic of propofol and remifentanil

INTERVENTIONS:
Drug: Pharmacokinetic of propofol and remifentanil — Pharmacokinetic of propofol and remifentanil in both population: Obese and non Obese patients

SUMMARY:
This prospective monocentric phamacokinetics study aims to compare plasmatic concentrations of Propofol and Remifentanil required to target a specific range of monitored anesthesia and analgesia during sus-mesocolic surgery in obese and non obese patients.

DETAILED DESCRIPTION:
Remifentanil and Propofol are administered intravenously as an opioid pain reliever and hypnotic pain reliever during anesthesia. Their advantages are numerous: short half-life allowing anesthesia and rapid awakening, little accumulation, allowing to adapt the level of anesthesia or sedation to each patient, few side effects.

Entropy° is an index derived from the electroencephalographic signal of patients, validated for the evaluation of the level of narcosis during general anesthesia.

ANI ° (nociception index analgesia) is an index using the ventilatory physiological variability of the sinus rhythm validated to monitor patient's analgesia during general anesthesia.

These non-invasive means of analgesia and sedation monitoring allows the clinician to ensure satisfactory levels of anesthesia by administering products at minimum effective doses.

The authors propose to determine whether, for a comparable target effect (analgesia and monitored sedation), plasmatic concentrations and administration rates of propofol and remifentanil necessary during general anesthesia for a comparable surgical stimulus are the same in populations of obese and non obese patients.

ELIGIBILITY:
Inclusion Criteria:

Obese patients group:

* Age ≥ 18 years old
* Severe and morbidly obese patients (35kg / m2≤IMC <55kg / m2).
* Patients undergoing general anesthesia for laparoscopic susmesocolic surgery (bariatric surgery or cholecystectomy).
* Patients who have given their consent in the manner described by the public health law of August 9, 2004.
* Patients benefiting from a Social Security scheme.

Group of non-obese patients:

* Age ≥ 18 years old
* Patients with normal weight or slightly overweight (19 <BMI <30).
* Patients receiving general anesthesia for laparoscopic susmesocolic surgery (cholecystectomy).
* Patients who have given their consent in the manner described by the public health law of August 9, 2004.
* Patients benefiting from a Social Security scheme.

Exclusion Criteria:

* Patient refusal
* Age <18 years old
* Protected adults and vulnerable persons
* Pace maker
* General anesthesia in the 24 hours preceding this surgery
* Proven or suspected dysautonomia
* Premedication by gabapentin Neurontin °
* Locoregional peri-medullary analgesia technique used concomitantly during the pre- and intraoperative period.
* Unbalanced dysrhythmic heart disease (AC / FA; extrasystoles; non-sinus rhythm)
* Pregnant or breastfeeding woman
* Intubation impossible planned
* Hypersensitivity to the products used
* Allergy to peanut or soy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of Propofol | 5 minutes after the insufflation of the pneumoperitoneum
  Plasma concentration of Propofol at different times during the maintenance phase of general anesthesia
Plasma concentration of Propofol | 5 minutes after completion of the gastric slice or ligation of the bile ducts
  Plasma concentration of Propofol at different times during the maintenance phase of general anesthesia
Plasma concentration of Propofol | At time of removing surgical specimen from the abdomen
  Plasma concentration of Propofol at different times during the maintenance phase of general anesthesia
Plasma concentration of Propofol | At the exsufflation of the pneumoperitoneum
  Plasma concentration of Propofol at different times during the maintenance phase of general anesthesia
Plasma concentration of Remifentanil | 5 minutes after the insufflation of the pneumoperitoneum
  Plasma concentration of Remifentanil at different times during the maintenance phase of general anesthesia
Plasma concentration of Remifentanil | 5 minutes after completion of the gastric slice or ligation of the bile ducts
  Plasma concentration of Remifentanil at different times during the maintenance phase of general anesthesia
Plasma concentration of Remifentanil | At time of removing surgical specimen from the abdomen
  Plasma concentration of Remifentanil at different times during the maintenance phase of general anesthesia
Plasma concentration of Remifentanil | At the exsufflation of the pneumoperitoneum
  Plasma concentration of Remifentanil at different times during the maintenance phase of general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Etienne Bazin, Pr, Principal Investigator — Service d'Anesthésie-Réanimation, Pôle Médecine Périopératoire - Hôpital Estaing, CHU de Clermont-Ferrand
Locations (1):
- Service d'Anesthésie-Réanimation, Pôle Médecine Périopératoire - Hôpital Estaing, CHU de Clermont-Ferrand, Clermont-Ferrand, Puy De Dôme, France